CLINICAL TRIAL: NCT03463187
Title: A Multi-Center, Randomized, Double-blind, Placebo-controlled, Multi-Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of SHR-1314 With Expanded Dose Finding in Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: Multi-Dose Study of SHR-1314 in Subjects With Moderate-to-severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1314-A201
Record Dates: First submitted 2018-01-22; First posted 2018-03-13 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Moderate-to-severe Chronic Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: PartA is a multiple dose escalating design in 3 sequential cohorts at 3 dose levels (80mg, 160mg, and 240mg) in plaque psoriasis subjects.
  Part B is a multiple dose, parallel-group design consisting of 4 treatment arms and 1 placebo arm to assess the efficacy and safety of s.c. injections of SHR-1314 in plaque psoriasis subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 80mg SHR-1314-Part A (Experimental): SHR-1314 80mg, subcutaneously
  Interventions: Biological: SHR-1314; Drug: Placebo
- 160mg SHR-1314-Part A (Experimental): SHR-1314 160mg, subcutaneously
  Interventions: Biological: SHR-1314; Drug: Placebo
- 240mg SHR-1314-Part A (Experimental): SHR-1314 240mg, subcutaneously
  Interventions: Biological: SHR-1314; Drug: Placebo
- 40mg SHR-1314 (Part B) (Experimental): SHR-1314 40mg, subcutaneously
  Interventions: Biological: SHR-1314
- 80mg SHR-1314 (Part B) (Experimental): SHR-1314 80mg, subcutaneously
  Interventions: Biological: SHR-1314
- 160mg SHR-1314 (Part B) (Experimental): SHR-1314 160mg, subcutaneously
  Interventions: Biological: SHR-1314
- 240mg SHR-1314 (Part B) (Experimental): SHR-1314 240mg, subcutaneously
  Interventions: Biological: SHR-1314
- SHR-1314 Placebo (Part B) (Experimental): SHR-1314 Placebo, subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: SHR-1314 — Administered subcutaneously
  Arms: 160mg SHR-1314 (Part B); 160mg SHR-1314-Part A; 240mg SHR-1314 (Part B); 240mg SHR-1314-Part A; 40mg SHR-1314 (Part B); 80mg SHR-1314 (Part B); 80mg SHR-1314-Part A
Drug: Placebo — Administered subcutaneously
  Arms: 160mg SHR-1314-Part A; 240mg SHR-1314-Part A; 80mg SHR-1314-Part A; SHR-1314 Placebo (Part B)

SUMMARY:
This is a multi-regional, randomized, double-blind, placebo-controlled, clinical trial to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of SHR-1314 in adults with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This study is a multiple dose escalating design to evaluate the safety, PK, and pharmacodynamics (PD) of multiple subcutaneous injections of SHR-1314. There are two parts in this study. The safety, PK, and PD will be evaluated in Part A, the dose escalation part. The efficacy and safety on different doses will be assessed in parallel-groups in Part B.

ELIGIBILITY:
Major Inclusion Criteria:

1. Provide written informed consent before any study assessment is performed.
2. Male or female at least 18 years of age at screening.
3. At the time of randomization, moderate to severe plaque psoriasis, defined by:

   * PASI score of 12 or greater and
   * PGA score of 3 or greater and
   * BSA affected by plaque-type psoriasis of 10% or greater.
4. Subject is a candidate for systemic psoriasis therapy and/or phototherapy and/or chemo phototherapy.

Major Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic, and guttate psoriasis) at screening.
2. Drug-induced psoriasis (i.e. new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) at randomization.
3. Active systemic infections (other than common cold) during the two weeks before randomization (e.g., hepatitis), or serious infections requiring hospitalization and/or intravenous injection of antibiotic treatment within eight weeks from randomization.
4. Presence of other skin conditions (e.g. skin infections, seborrheic dermatitis) that in the judgement of the Investigator could interfere with assessment of psoriasis.
5. History of inflammatory bowel disease or have other ongoing active autoimmune diseases.
6. At screening, history or symptoms of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
7. History of depression and/or suicidal ideation or behavior which in the opinion of the Investigator, makes the subject unsuitable for clinical study participation.
8. Any severe, progressive or uncontrolled medical condition at randomization that in the judgement of the Investigator prevents the subject from participating in the study.
9. Have a known allergy or hypersensitivity to any biologic therapy at screening that would pose an unacceptable risk to the subject if participating in this study.
10. Concurrent or recent use of psoriasis treatments/ medications.
11. Are currently enrolled in, or discontinued from a clinical trial involving an Investigational product (IP) within the last 4 weeks or at least 5 half-lives of the last dosing prior to randomization, whichever is longer; or concurrently enrolled (at randomization) in any other trials.
12. Have had a live attenuated vaccination within 12 weeks before randomization, or intend to have a live attenuated vaccination during the course of the study, or have participated in a vaccine clinical trial within 12 weeks prior to randomization.
13. Have evidence of positive test for hepatitis B, hepatitis C antibody, or human immunodeficiency virus (HIV) antibodies.

    A positive test for hepatitis B is defined as 1) positive for hepatitis B surface antigen [HBsAg], or 2) positive for anti-hepatitis B core antibody [HBcAb+] but negative for hepatitis B surface antibody [HBsAb-].
14. History or evidence of active or latent tuberculosis at screening.
15. Have laboratory test values that are considered clinically significant at screening that, in the opinion of the Investigator, pose an unacceptable risk to the subject if participating in the study or of interfering with the interpretation of data.
16. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test at screening or Day 0.
17. Females of child bearing potential (defined as all females physiologically capable of becoming pregnant) and males who are unwilling or unable to use highly effective contraception during the study and 20 weeks after the last administration of investigational product (anticipated 5 half-lives).
18. History of alcohol or illicit drug abuse within the year prior to screening.
19. Are unwilling or unable to maintain their normal pattern of alcohol, caffeine, smoking, and exercise from the start to the end of the study.
20. Have any other condition that precludes the subject from following and completing the protocol, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Clinically Significant Events (Part A) | From baseline through 24 weeks
  Clinically significant events were defined as abnormal laboratory values and/or adverse events that are related to treatment
Pharmacokinetics (PK) of SHR-1314 (Part A) | From baseline through 24 weeks
  Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Pharmacokinetics (PK) of SHR-1314 (Part A) | From baseline through 24 weeks
  Observed Maximum Serum Concentration Following Drug Administration (Cmax)
Percentage of Participants With Anti-SHR-1314 Antibodies (Part A) | From baseline through 24 weeks
  Percentage of participants with treatment-emergent positive anti-SHR-1314 antibodies was summarized by treatment group. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-SHR-1314 antibodies / number of evaluable participants * 100%.
Percentage of subjects who achieve Psoriasis Area Severity Index (PASI) score 75 (Part B) | From baseline through 12 weeks
  Percentage of subjects who achieve at least 75% improvement in the PASI (PASI 75)

SECONDARY OUTCOMES:
Psoriasis Area Severity Index (PASI) score | From baseline through 24 weeks (Part A) or 36 weeks (Part B)
  PASI combines the extent of body surface involvement in 4 anatomical regions(head,trunk,arms,and legs).For each region the percent area of skin involved was estimated from 0(0%) to 6(90%-100%) and severity was estimated by clinical signs of erythema,induration and scaling with a scores range from 0(none) to 4(very severe).Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as:sum of severity parameters for each region*area score*weighing factor (head[0.1],upper limbs[0.2],trunk[0.3],lower limbs [0.4]).Overall scores range from 0(no psoriasis) to 72(most severe disease). Percent change from baseline in PASI score over time will be evaluated.
Physician's Global Assessment (PGA) of 0 or 1 achievement | From baseline through 24 weeks (Part A) or 36 weeks (Part B)
  The PGA of psoriasis is scored on a 6-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 6-point severity scale (0 [clear] to 5 [severe]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=moderate to severe; 5 = severe). Proportion of subjects achieving PGA response of 0 or 1 over time will be evaluated. PGA response of 0 or 1 is defined as a PGA score of 0 (clear) or 1 (almost clear) and an improvement of at least 2 points on the PGA scale from baseline.
Change of dermatology life quality index (DLQI) score | From baseline up to 12 weeks (Part A) or 36 weeks (Part B)
  Change from baseline in DLQI over time. This DLQI is a 10-question patient administered questionnaire that covers six quality of life domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment, with total scores ranging from 0-30 (less to more impairment)
Change from baseline in Body Surface Area (BSA) | From baseline through 12 weeks (Part A) or (Part B)
  Change from baseline in the BSA affected by psoriasis over time.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Revival Research, Doral, Florida
  - Indago Research and Health Center - Emergency Medicine, Hialeah, Florida
  - Great Lakes Clinical Trials LLC, Chicago, Illinois
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
- Australia (4):
  - St George Dermatology and Skin Cancer Centre - Dermatology, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Sinclair Dermatology - Dermatology, East Melbourne, Victoria
- Shanghai Huanshan Hospital Fudan University-Dermatology, Shanghai, China

REFERENCES:
- [Derived] Zhang C, Yan K, Diao Q, Guo Q, Jin H, Yang S, Chen X, Lei T, Wu J, Yu H, Zheng M, Gao X, Sinclair R, Zhu Y, Xu Q, Xu J. A multicenter, randomized, double-blinded, placebo-controlled, dose-ranging study evaluating the efficacy and safety of vunakizumab in patients with moderate-to-severe plaque psoriasis. J Am Acad Dermatol. 2022 Jul;87(1):95-102. doi: 10.1016/j.jaad.2022.01.005. Epub 2022 Jan 10. PMID 35026342